CLINICAL TRIAL: NCT05126355
Title: Effectiveness of the On the Move Group Exercise Program to Improve Mobility in Community-dwelling Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jennifer S. Brach, Professor and Associate Dean for Faculty Affairs and Development, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY21070206; R01AG071520 (NIH)
Record Dates: First submitted 2021-11-01; First posted 2021-11-19 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Mobility Limitation
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- On the Move (Experimental): On the Move group exercise program to improve walking. Delivered twice per week for 12 weeks.
  Interventions: Behavioral: On the Move group exercise
- On the Move - Delayed (Other): Individuals in this arm will be placed on a wait-list for 12 weeks and will receive no intervention during this time. At the end of the 12 weeks they will receive the On the Move group exercise program. This is a wait-list control group.
  Interventions: Behavioral: On the Move group exercise

INTERVENTIONS:
Behavioral: On the Move group exercise — The OTM exercise program is a group-based program led by a certified OTM instructor. The frequency and duration of OTM is 50 minutes, twice weekly for 12 weeks for a total of 24 classes. The OTM exercise program is based on principles of motor learning that enhance smooth and automatic movement control. The program contains a warm-up (5 minutes), stepping patterns (15 minutes), walking patterns (15 minutes), strengthening exercises (10 minutes), and cool-down exercises (5 minutes). The warm-up and cool down contain gentle range of motion exercises and stretches for the lower extremities and trunk. Considered essential components, the stepping and walking patterns are progressively more difficult, goal-oriented patterns that promote the timing and coordination of stepping integrated with the phases of the gait cycle.

SUMMARY:
The purpose of this study is to test the effectiveness of On the Move (OTM) in terms of improving mobility among 502 older adults in 44 senior community centers and to evaluate intervention fidelity, including adherence and competence, and the impact of organizational, instructor, and participant level factors on intervention fidelity.

DETAILED DESCRIPTION:
The investigators will conduct a Hybrid I trial, blending effectiveness and implementation research aims to: test the effectiveness of OTM, evaluate intervention fidelity, and determine the extent intervention fidelity moderates intervention effectiveness. The investigators will evaluate the effects of OTM taught by community instructors for improving mobility among 502 older adults in 44 community centers using a cluster randomized design with a delayed intervention control arm. Intervention fidelity will be assessed by instructor self-report (intervention diaries) and observation (fidelity checklist). Organizational, instructor, and participant level factors which may impact fidelity will be assessed via standard instruments, focus groups and interviews.

Specific Aims are as follows:

Aim 1: Establish the effectiveness of OTM on improvements in walking ability and post-intervention persistence of benefits.

Rationale: OTM delivered by research staff is effective. Establishing the effectiveness of OTM delivered by community instructors is necessary before wide-scale implementation.

Hypothesis: Compared to a randomized control group followed for 12 weeks, the OTM group will have greater gains in gait speed (primary outcome) and self-reported mobility at 12 and 24 weeks of follow-up.

Aim 2: Assess intervention fidelity (measures of adherence and competence) and identify the impact of organizational, instructor, and participant level factors on intervention fidelity.

Rationale: To inform future implementation efforts, it is critical to measure intervention fidelity and to identify factors associated with fidelity.

Hypothesis: Organizational, instructor, and participant level factors will impact fidelity. For example, instructors who utilize greater facilitation strategies will have higher fidelity, poor organizational acceptance of the program will be related to lower fidelity, and fewer organizational resources will lead to lower fidelity.

Aim 3: Determine the extent to which intervention fidelity, measured by adherence and competence, moderates the effectiveness of OTM.

Rationale: Intervention fidelity may influence the effectiveness of OTM. Understanding the consequences of differing levels of intervention fidelity on effectiveness will inform future implementation efforts.

Hypothesis: Higher fidelity will be associated with greater mobility gains, and there may be critical fidelity thresholds.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* attend the senior center
* can ambulate household distances independently
* can participate in group exercise classes

Exclusion Criteria:

* impaired cognition (unable to understand consent process)
* plans to leave the area for an extended period of time
* any acute or unstable illness or medical condition

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Gait speed | 12 weeks
  The time it take the subject to walk 4 meters and their usual walking speed. Recorded as m/s. Faster speeds indicate better mobility.
Gait speed | 24 weeks
  The time it take the subject to walk 4 meters and their usual walking speed. Recorded as m/s. Faster speeds indicate better mobility.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) mobility | 12 weeks
  The Patient-Reported Outcomes Measurement Information System - mobility measure is 15 item scale to assess self-reported perceptions of mobility. A single mobility score is obtained from the short form, with higher scores indicating better mobility.
Patient-Reported Outcomes Measurement Information System (PROMIS) mobility | 24 weeks
  The Patient-Reported Outcomes Measurement Information System - mobility measure is 15 item scale to assess self-reported perceptions of mobility. A single mobility score is obtained from the short form, with higher scores indicating better mobility.
Participant Satisfaction | immediately post intervention
  Participant satisfaction will be assessed using a survey that includes five items measured on a Likert scale and three yes/no questions. The Likert items assess degree of satisfaction with various components of the exercise program (i.e. the exercises, instructor, music, space, and the overall program). The yes/no questions assess if the program met the participants' expectations, if they feel they benefited from the program, and if they would recommend the program to others.

OTHER OUTCOMES:
Adherence - Content | Throughout the 12 week intervention
  We have identified the essential components of OTM. Inclusion of essential components will be determined from exercise class logs. OTM instructors will be required to keep a log of time spent on each program component in each class, for each of the 24 classes. We will review the logs and determine if the essential components (warm-up, walking, stepping patterns, strengthening exercises and cool-down) are included in each of the classes. For each of the classes offered, instructors will be classified as being fully adherent, adherent to core components only, or non-adherent.
Adherence - Dose of exposure classes offered | Throughout the 12 week intervention
  Dose of exposure classes offered will be quantified as number of classes offered by the community center (0-24). Each community center is required to document when exercise classes are offered. The investigators will obtain this information directly from the community center records. A greater number of classes is better.
Adherence - Dose of exposure, weeks of exercise | Throughout the 12 week intervention
  Dose of exposure, weeks of exercise will be quantified as the number of weeks the exercise classes are offered (0-12). Each community center is required to document when exercise classes are offered. The investigators will obtain this information directly from the community center records. A greater number of weeks is better.
Adherence - Dose of exposure, participant level. | Throughout the 12 week intervention
  Dose of exposure at the participant level will be quantified as the number of classes each participant attends, 0-24. The instructor will keep a class log of each session to record attendance. A greater number of classes is better.
Competence - Quality of delivery | Throughout the 12 week intervention
  The content experts will use a standardized checklist to document if the instructor is delivering the program with adequate skill. The checklist includes 20 items such as appropriately demonstrating exercises, modifying the exercises as needed, and progressing exercises appropriately. Competence will be quantified by the total number of items present on the checklist; scores will range from 0-20.
Adaptations | Throughout the 12 week intervention.
  Adaptations will be recorded, defined and classified using the Framework for Reporting Adaptations and Modifications-Expanded (FRAME).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Brach, PhD, PT, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data may be shared. Because the human subjects included in the project could potentially be identified, given the relatively limited geographic distribution of these subjects, investigators requesting data will be required to sign a data sharing agreement. For external requests, the agreement will be executed through the University's Office of Research; and for internal requests, through email.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data sets will be available at the time the primary paper is accepted for publication or at 2 years after the last participant is followed whichever comes first.
Access Criteria: Data will be available by secure transfer to investigators who complete a data sharing agreement for data from this project. The sharable data will be archived at the study's home site and will be available for sharing by submitting a request to the PI. Once a request is approved by the PI and the requester agrees to the conditions for data use, the data will be transferred.